CLINICAL TRIAL: NCT00960648
Title: EXCELLENT (Efficacy of Xience/Promus Versus Cypher in rEducing Late Loss After stENTing) Registry
Brief Title: Registry to Evaluate Efficacy of Xience/Promus Versus Cypher in Reducing Late Loss After Stenting
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Abbott (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Hyo-SOO Kim, MD, PhD, Seoul National University Hospital
Other Study IDs: EXCELLENT-REGISTRY
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Artery Disease
Keywords: Everolimus; Sirolimus; Drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Xience/Promus: Active prospective registration of patients receiving everolimus eluting stent
  Interventions: Device: Xience/Promus
- Cypher: Retrospective historical controls that received sirolimus-eluting stent
  Interventions: Device: Cypher

INTERVENTIONS:
Device: Xience/Promus — Active prospective registration of patients receiving everolimus-eluting stent
  Other Names: EES
  Groups: Xience/Promus
Device: Cypher — Retrospective historical controls that received sirolimus-eluting stent
  Other Names: SES
  Groups: Cypher

SUMMARY:
The objective of this study is to evaluate the safety and long-term effectiveness of coronary stenting with the everolimus-eluting stent (EES) and to determine clinical device and procedural success during commercial use of EES in the real world.

The investigators will compare EES (Xience/Promus, prospective arm) with sirolimus-eluting stent (SES, Cypher, retrospective arm).

ELIGIBILITY:
Inclusion Criteria:

* The patient agrees to participate in this study by signing the informed consent form.
* Alternatively, a legally authorized patient representative may agree to the patient's participation in this study and sign the informed consent form.

Exclusion Criteria:

* There are no exclusion criteria for this registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 4000 patients derived from a population of patients receiving percutaneous coronary intervention for ischemic heart disease will be enrolled in the present registry.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (composite of cardiac death, non-fatal MI, target lesion revascularization) | 12 months

SECONDARY OUTCOMES:
In-stent & In-segment Late Loss | 9 months
Stent Thrombosis | 1 year
Target Vessel Failure (composite of cardiac death, MI, and TVR) | 12 months
Any death, cardiac death, MI, TLR, TVR | 1 year
Composite rate of cardiac death and any MI | 1 year
Composite rate of all death and any MI | 1 year
Composite rate of all death, any MI (Q-wave and non Q-wave) and any repeat revascularization | 1 year
Compliance and therapy interruptions with prescribed adjunctive antiplatelet therapy | 1 year
Clinical device and procedural success | During the health care facility stay

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD,PhD, Study Chair — Seoul National University Hospital
Locations (18):
- South Korea (18):
  - Dankook University Hospital, Cheonan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Kwangju Veterans Hospital, Gwangju
  - Chonbuk National University Hospital, Iksan
  - Wonkwang University Hospital, Iksan
  - Inje University Ilsan Paik Hospital, Ilsan
  - Gachon Kil Medical Center, Inchon
  - Chungbuk National University Hospital, Jeonju
  - Presbyterian Medical Center, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Inje University Pusan Paik Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Gangnam Severance Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Medical Center, Seoul
  - St. Carollo Hospital, Suncheon